CLINICAL TRIAL: NCT05753046
Title: Perioperative Laparoscopic Transversus Abdominis Plane Block During Robotic Assisted Laparoscopic Radical Prostatectomy for Improvement in Postoperative Pain
Brief Title: Laparoscopic TAP Block During Robotic Assisted Laparoscopic Radical Prostatectomy for Improvement in Postoperative Pain
Acronym: TAPBlock
Status: Enrolling by invitation | Phase: Phase 4 | Type: Interventional
Sponsor: Corewell Health East (Other)
Responsible Party: Principal Investigator, S Mohammad Jafri, Urologist, Corewell Health East
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 2022-235
Record Dates: First submitted 2023-02-21; First posted 2023-03-03 (Actual); Last update posted 2025-04-27 (Actual); Status verified 2025-04

CONDITIONS: Prostate Cancer
Keywords: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Intervention Model Description: Patients who meet all eligibility criteria will be enrolled in the study and randomized (1:1) to receive either early or late TAP block. The subject and biostatistician will be blinded to the group allocation throughout the study. Research staff responsible for obtaining consent. To maintain the blind, initial analysis of the data performed by the biostatistician will not include group assignment.
Who Masked: Participant, Outcomes Assessor
Masking Description: Patients will be sedated for the procedure and unaware of when the TAP block is administered.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Early TAP Block (Experimental): For treatment delivery, subjects will receive 60 mL of 0.25 percent ropivacaine with 4 mg of dexamethasone at the initiation of the procedure (immediately following placement of the robotic / laparoscopic camera port).
  Interventions: Drug: Early TAP Block
- Late TAP Block (Experimental): For treatment delivery, subjects will receive 60 mL of 0.25 percent ropivacaine with 4 mg of dexamethasone either at the conclusion of the procedure (immediately preceding removal of the robotic / laparoscopic camera port).
  Interventions: Drug: Late TAP Block

INTERVENTIONS:
Drug: Early TAP Block — For treatment delivery, subjects will receive 60 mL of 0.25 percent ropivacaine with 4 mg of dexamethasone at the initiation of the procedure (immediately following placement of the robotic / laparoscopic camera port). The TAP block will be performed with 15 mL 2 finger breadths subcostal at the mid-clavicular line and then 15 mL at the level of the umbilicus along the mid-axillary line on each side. Laparoscopic / robotic camera will be used as a visual aid to confirm positioning between the internal oblique and transversus abdominis muscles for the goal of pain relief.
  Other Names: Initiation of procedure
  Arms: Early TAP Block
Drug: Late TAP Block — For treatment delivery, subjects will receive 60 mL of 0.25 percent ropivacaine with 4 mg of dexamethasone at the conclusion of the procedure (immediately proceeding removal of the robotic / laparoscopic camera port). The TAP block will be performed with 15 mL 2 finger breadths subcostal at the mid-clavicular line and then 15 mL at the level of the umbilicus along the mid-axillary line on each side. Laparoscopic / robotic camera will be used as a visual aid to confirm positioning between the internal oblique and transversus abdominis muscles for the goal of pain relief.
  Other Names: Conclusion of procedure
  Arms: Late TAP Block

SUMMARY:
Determine the impact of a laparoscopic-guided transversus abdominis plane (TAP) block timing (at initiation or conclusion of procedure) on the postoperative pain experience in patients following robot assisted laparoscopic radical prostatectomy (RALP).

DETAILED DESCRIPTION:
TAP block involves the use of a local anesthetic agent injected between the internal oblique and transversus abdominis muscles for the goal of pain relief. Often times these are performed under ultrasound guidance by the anesthesiology team preoperatively. The idea behind this is to provide a neurologic block to the sensory nerve fibers supplying the anterior abdominal wall, between the internal oblique and transversus abdominis muscles. More recently, this technique has been investigated in the setting of robot-assisted laparoscopic radical prostatectomy (RALP) with promising results. There is a lack of data comparing the benefits of the timing of TAP block, and whether performing this at the initiation versus conclusion of the case provides superior results

This is a prospective, randomized controlled trial of subjects undergoing early versus late TAP block for the management of postoperative pain following RALP. Subjects will be recruited through physician referral from private Urology offices. Potential subjects (patients scheduled for RALP procedure) will be approached by the study doctor prior to surgery, either in the study doctor's office or in the pre-operative area.

Subjects who meet all the eligibility criteria will be enrolled in the study and randomized (1:1) to receive early or late surgeon performed laparoscopic TAP block. Each patient will only receive one treatment (TAP block) either at the initiation or conclusion of his procedure.

For treatment delivery, subjects will receive 60 mL of 0.25 percent ropivacaine with 4 mg of dexamethasone either at the initiation of the procedure (immediately following placement of the robotic / laparoscopic camera port) or at the conclusion of the procedure (immediately proceeding removal of the robotic / laparoscopic camera port). Study doctors will use laparoscopic / robotic camera visual aid to confirm positioning between the internal oblique and transversus abdominis muscles for the goal of pain relief.

ELIGIBILITY:
Inclusion Criteria:

1. Able to read, understand, and provide written, dated, informed consent prior to screening, complete study form(s) independently, comply with study protocol, and communicate with study personnel about clinically important information.
2. Men ≥ 18 years of age.
3. Pathologically confirmed diagnosis of prostate cancer
4. Scheduled for routine RALP

Exclusion Criteria:

1. Chronic opioid use (daily for >3 months)
2. Weight <40 kilograms
3. Any condition that causes a lack of normal sensation to the abdomen or pelvis
4. Current or history of any physical condition that, in the investigator's opinion, might put the subject at risk or interfere with study results interpretation

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Men with pathologically confirmed diagnosis of prostate cancer
Enrollment: 94 (Estimated)
Dates: Start 2024-02-19 (Actual); Primary Completion 2028-08 (Estimated); Study Completion 2029-08 (Estimated)

PRIMARY OUTCOMES:
Compare laparoscopic-guided TAP block timing (at initiation "early" or conclusion "late" of procedure) on the postoperative pain levels reported in patients following robot assisted laparoscopic radical prostatectomy (RALP). | 24 hours after RALP
  Comparison of patient reported pain scales, based on a score from 0 to 10. Where 0 is no pain and 10 is the worst pain.

SECONDARY OUTCOMES:
Compare the effects of TAP Block timing on total opioid consumption | 7 days after RALP with TAP Block
  Total opioid consumption will be calculated in morphine equivalent dose (MED).
Compare the effects of TAP Block timing on hospital length of stay | 7 days after RALP with TAP Block
  Total number of days hospitalized from day of procedure to day of discharge home. Reported in number of days.
Compare the effects of TAP Block timing on return of bowel function | 7 days after RALP with TAP Block
  When the patient reports the occurrence of the first bowel movement following the procedure. Reported in number of days.
Compare the effects of TAP Block timing on postoperative nausea/vomiting | 7 days after RALP with TAP Block
  Total number of patient reported occurrences of nausea/vomiting documented in the medical record.
Compare the effects of TAP Block timing on ambulation | 7 days after RALP with TAP Block
  The time in hours reported after the first recorded ambulation post procedure in the medical record.
Compare the effects of TAP Block timing on readmission for pain | 7 days after RALP with TAP Block
  The time in days following discharge to readmission with the rationale for admission noted as pain.
Compare the safety and tolerability of laparoscopic TAP block. | 7 days after RALP with TAP Block
  Safety and tolerability of laparoscopic TAP Block will be assessed in relation to the incidence of adverse events reported.

CONTACTS AND LOCATIONS:
Overall Officials: S. Mohammad Jafri, MD, Principal Investigator — Corewell Health William Beaumont University Hospital
Locations (1):
- Corewell Health William Beaumont University Hospital, Royal Oak, Michigan, United States

IPD SHARING:
Plan to Share IPD: No